CLINICAL TRIAL: NCT07273409
Title: PANcreatic Neuroendocrine Tumour - Optimal Surgical Debulking Or Not (PANTODON). A Prospective, Two Armed, Parallel, Randomised, Controlled International Multicentre Study on WHO Grade 1-2, Stage 4 Pancreatic NET
Brief Title: Pancreatic Neuroendocrine Tumour - Optimal Surgical Debulking or Not
Acronym: PANTODON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala Clinical Research Center, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PANTODON/2025
Record Dates: First submitted 2025-09-24; First posted 2025-12-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Neuroendocrine Tumor
Keywords: Pan-NET; Stage 4; Debulking surgery; Non-functional Pan-NET; GI-WHO grade 1-2 Pan-NET
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Prospective, two armed, parallel, randomised, controlled, international multi-centre study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical group (Experimental): Debulking surgery followed by oncologic treatment according to standard routine. Further debulking surgery or ablation may be continued during follow-up to reduce tumour load.
  Interventions: Procedure: Debulking surgery
- Non-surgical group (No Intervention): Oncologic treatment alone. No surgical or thermal ablative treatments will be planned after randomisation. Any surgical or ablative procedure for pan-NET that is performed after randomisation in the Non-surgical group is considered as a protocol deviation. However, such procedures may be carried out if clinically indicated and no other equivalent or better oncological options for treatment are available. The surgery is then documented as oncological treatment in eCRF and the subject will continue follow-up in the study.

INTERVENTIONS:
Procedure: Debulking surgery — All subjects are divided into STRATUM 1 and STRATUM 2 prior to randomisation.
  For subjects in STRATUM 1, the surgical resection, alone or in combination with ablative procedures, aim to achieve at least 70% debulking of the total tumour volume, with acceptable risk and acceptable functional liver remnant (FLR).
  For subjects in STRATUM 2 the aim is to resect or ablate all FluDeoxyGlucose-Positron emission tomography (FDG-PET) avid disease with acceptable risk and acceptable FLR.
  Arms: Surgical group

SUMMARY:
Pancreatic neuroendocrine tumours (pan-NETs) are neoplasms arising from the endocrine cells of the pancreas. Although pan-NET are quite rare, the incidence is on the rise and together with other abdominal neuroendocrine tumours an approximate incidence in Sweden would be 850 patients per year extrapolating from Norwegian data. Pan-NET are divided into symptomatic hormone producing tumours (such as insulinomas/glucagonomas/VIPomas) or non-functioning tumours that often are asymptomatic. As early symptoms often are lacking in non-functioning-pan-NET, many patients present with distant metastases and are thus beyond a curative surgical approach at the time of diagnosis. Metastatic non-functioning pan-NETs present a significant challenge and the optimal management remains a subject of debate.

This is a prospective, two armed, parallel, randomised, controlled, international multi-centre study, aiming to investigate if a near-total tumour debulking (intervention) in metastatic (stage 4) GI-WHO grade 1-2 pan- NET, with or without oncologic treatment, is superior to oncologic treatment alone (control), with regards to overall survival, health-related quality of life, participant performance status, time until hospitalisation, adverse event characteristics and cost in the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* Pan- NET, ENETS/AJCC stage 4 determined by CT or PET/CT
* Primary tumour or metastases confirmed as Pancreatic NET GI-WHO grade 1-2 pan-NET by histology or cytology
* Age ≥ 18 years
* Written informed consent obtained

Exclusion Criteria:

* Subject not fit for surgery due to comorbidity or advanced age (reason to be specified)
* Risk of surgery deemed too high by MDT or Surgeon (reason to be specified)
* Previous surgery for pan-NET.
* Hormonal symptoms caused by a functional pan-NET, not controllable by medical therapy, indicating debulking surgery.
* Previously included in the current study.
* Pregnancy
* The study subject does not fit into either STRATA: a) STRATUM 1: Less than 70% of the total tumour volume can be debulked, b) STRATUM 2: no FDG-PET avid disease is observed OR all (100%) FDG-PET avid tumour is not resectable.
* Other reason in the opinion of the Principal Investigator (reason to be specified).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2033-05-31 (Estimated); Study Completion 2033-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Five years or until death.
  Time from randomisation to death.

SECONDARY OUTCOMES:
Health economics | Until end of trial.
  Estimation of total health economic costs for hospitalisation, ICU stay, and treatments given for the pan-NET disease in each group during follow-up.
Health-related quality of life | The questionnaire will be filled in by the study subject before randomisation, at 3 months (+/2weeks), 6 months, and at 1, 2, 3, 4 and 5 years (+/4weeks) after randomisation.
  Data on health-related quality of life will be gathered with the EORTC Core Quality of Life questionnaire (EORTC QLQ-C30). The questionnaire is designed to measure cancer subjects' physical, psychological and social functions. It is composed of multi-item scales and single items.
Performance status | Assessed at screening, at 3 months (+/2weeks), 6 months, and at 1, 2, 3, 4 and 5 years (+/4weeks) after randomisation.
  Performance status is measured using the Karnofsky performance status scale The scale ranges from 100 to 0, with higher scores indicating better functional status.
Days out of hospital | Assessed at 3 months (+/2weeks), 6 months, and at 1, 2, 3, 4 and 5 years (+/4weeks) after randomisation.
  Total number of days alive outside hospital.
Days out of intensive care unit | Assessed at 1 and 5 years.
  Total number of days alive outside intensive care unit.
Adverse events | From randomisation until the end of the study period.
  Severe, life threatening and fatal adverse events possibly or probably related to pan-NET treatment during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Olov Norlén, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (4):
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided